CLINICAL TRIAL: NCT06014307
Title: SWAP-MEAT (Study With Appetizing Plant-Food, Meat Eating Alternatives Trial) Athlete for MC-URC (Menus of Change University Research Collaborative): Three Diets on Athletic Performance
Brief Title: SWAP-MEAT With Athletes for MC-URC: Three Diets on Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 69487
Record Dates: First submitted 2023-08-23; First posted 2023-08-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Health Behavior
Keywords: muscular strength; endurance; plant-based diets; meat alternatives; omnivore diets
MeSH Terms: conditions — Health Behavior | interventions — polybutyl methacrylate

STUDY DESIGN:
Intervention Model Description: SWAP-MEAT Athlete is a randomized crossover trial in which 10 recreational runners and 10 recreational resistance trainers are assigned to one of six possible diet orders. Each diet order contains three phases for 4 to 6 weeks each (4 weeks for universities on the quarter system; 6 weeks for universities on the semester system) -Animal, Plant-Based Meat Alternatives (PBMA), and Whole Food Plant-Based (WFPB)-in random order.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-Based Meat Alternatives (PBMA) (Experimental): Up to 2 servings per day of plant-based meat alternatives (Beyond Beef, Impossible Burger, Gardein Chick'n) OR as many plant-based meat alternative servings as available per day in the dining halls.
  Interventions: Behavioral: Diet order: PBMA, Animal; Behavioral: Diet order: Animal, PBMA
- Animal (Experimental): 2 servings/day of traditional meat products (beef burger, pork, chicken)
  Interventions: Behavioral: Diet order: PBMA, Animal; Behavioral: Diet order: Animal, PBMA

INTERVENTIONS:
Behavioral: Diet order: PBMA, Animal — Participants will follow the PBMA, and Animal diets (in this order) for 4-6 weeks each.
Behavioral: Diet order: Animal, PBMA — Participants will follow the Animal, and PBMA diets (in this order) for 4-6 weeks each.

SUMMARY:
This study aims to investigate the impact of two plant-based diets-whole food plant-based (WFPB) and plant-based meat alternatives (PBMA)-vs. an omnivorous diet (Animal) on endurance and muscular strength in recreational athletes.

DETAILED DESCRIPTION:
The SWAP-MEAT study compared the impact of consuming diets containing animal meat (primarily beef and pork) vs. plant-based alternative meats (Beyond Meat products) on health risk factors, cardiometabolic risk factors, and the gut microbiome in generally healthy adults. The SWAP-MEAT Athlete pilot study explored the impact of these diets on athletic performance instead of health biomarkers and cardiovascular disease.

The purpose of this study is to replicate the pilot study with the exception of using undergraduate students who have access to Stanford dining halls, rather than graduate students who have to buy and prepare their own food. It will be a 2x4-6 week randomized crossover trial that contains two arms: animal meat and plant-based alternative meat. Generally healthy recreational athletes will be recruited and complete athletic performance field tests at the end of each diet in order to assess athletic performance outcomes. From the SWAP-MEAT: Athlete pilot study, the investigators can attest to the feasibility of the trial and have justification for conducting this larger study.

This study will aim to focus on BIPOC (Black, Indigenous, People of Color) undergraduate students. By doing so, the investigators can gain a better understanding of the potential barriers and challenges to their adoption in diverse populations, for example, understanding of how cultural differences influence dietary choices and preconceptions about plant-based diets and animal protein alternatives. This study aims to address these limitations and provide valuable insights into the effectiveness of plant-based diets for recreational athletes, as well as potential barriers and challenges to their adoption in diverse populations.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy omnivorous adults between 18 and 35 years of age who report typically consuming at least 1 serving of meat per day and are willing to consume ~2 servings per day of animal meat, plant-based meat alternatives, and whole-food plant proteins.
* Participants will have been consistent recreational runners or weightlifters (3-4 times per week) for at least the prior 1 year, and currently run or lift 3-4 times per week.
* Runners will engage in at least 150 minutes of moderate-to-vigorous aerobic activity or 75 minutes of vigorous activity per week. All participants will have habitually consumed an omnivorous diet for at least months.
* Participants will have self-reported good health and BMI 18.5-30.0.
* Participants must be able to commit to running or resistance training at least 3-4 times per week for the duration of the study.
* Participants will be on a Stanford meal plan which allows them access to the nine dining halls on the Stanford campus.

Exclusion Criteria:

* Individuals who have participated in any restrictive diet within the last month, have any known nutrient intolerances, have orthopedic limitations, are participating in any other physical activity or diet study;
* Individuals consuming any performance-enhancing drugs or medications known to interfere with athletic performance;
* Individuals who have a chronic disease or eating disorder, are currently pregnant or intend to become pregnant in the next three months, or have an intent to compete in any physical activity competition within the next 3 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Cooper 12-Minute Timed Run Test (Runners) | Baseline, Week 4 or Week 6
  Change from baseline in distance covered on a 12-minute timed run after each diet phase
Composite Machine Strength Index (Resistance Trainers) | Baseline, Week 4 or Week 6
  Change from baseline in composite machine strength index (sum of 3-rep max chest press, leg press, biceps curls, and lat pull-down) after each diet phase

SECONDARY OUTCOMES:
Dietary intake and adherence | Baseline, Week 4 or Week 6
  Nutrient composition of each diet and adherence to diet in servings of protein source consumed per week, via weekly dietary logs.
Diet satisfaction | Baseline, Week 4 or Week 6
  Score on Food Acceptability Questionnaire, measuring taste, appeal, and overall diet satisfaction, after each diet. We used the "Food Acceptability Questionnaire", with a minimum value of 1 and a maximum value of 7. A higher score indicates better food acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (5):
- United States (4):
  - UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Rutgers University, New Brunswick, New Jersey
  - Vanderbilt University, Nashville, Tennessee
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crimarco A, Springfield S, Petlura C, Streaty T, Cunanan K, Lee J, Fielding-Singh P, Carter MM, Topf MA, Wastyk HC, Sonnenburg ED, Sonnenburg JL, Gardner CD. A randomized crossover trial on the effect of plant-based compared with animal-based meat on trimethylamine-N-oxide and cardiovascular disease risk factors in generally healthy adults: Study With Appetizing Plantfood-Meat Eating Alternative Trial (SWAP-MEAT). Am J Clin Nutr. 2020 Nov 11;112(5):1188-1199. doi: 10.1093/ajcn/nqaa203. PMID 32780794
- [Background] Roberts AK, Busque V, Robinson JL, Landry MJ, Gardner CD. SWAP-MEAT Athlete (study with appetizing plant-food, meat eating alternatives trial) - investigating the impact of three different diets on recreational athletic performance: a randomized crossover trial. Nutr J. 2022 Nov 16;21(1):69. doi: 10.1186/s12937-022-00820-x. PMID 36384651